CLINICAL TRIAL: NCT06868030
Title: Efficacy and Safety of Conventional Symptomatic Drugs Combined with Lencanizumab in the Treatment of Early Alzheimer's Disease: a Multicenter, Prospective, Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Liu Huayan, Neurology department, First Hospital of China Medical University
Other Study IDs: LiuHuayan
Record Dates: First submitted 2025-01-26; First posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-01

CONDITIONS: Alzheimer's Disease; MCI-AD, Early Stage Alzheimer's Disease
Keywords: Alzheimer disease; MCI-AD, early stage Alzheimer's disease; lencanizumab; treatment
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples and cerebrospinal fluid samples stored at -80℃
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Combination treatment group: no less than 60 early AD patients (MCI-AD and mild AD) were selected from 10 centers from January 2025 to June 2025. The AD diagnosis met the diagnostic criteria for dementia described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R), using the 2011 NIA-AA criteria for AD. The MCI diagnosis met the MCI diagnostic criteria for the 2004 Peterson.
- Conventional symptomatic treatment group: no less than 60 early AD patients (MCI-AD and mild AD) were selected from 20 centers from January 2025 to June 2024. The AD diagnosis met the diagnostic criteria for dementia described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R), using the 2011 NIA-AA criteria for AD. The MCI diagnosis met the MCI diagnostic criteria for the 2004 Peterson.

SUMMARY:
According to the World Health Organization, China will become the "oldest" country in the world by 2050, with 35 percent of the elderly population. At present, in the Chinese population of 60 years old, there are about 15.07 million dementia patients (about 6.0%), about 9.83 million Alzheimer's disease (AD) patients (about 3.9%), and about 38.77 million mild cognitive impairment (Mild cognitive impairment, MCI) patients (about 15.5%). A sharp increase in older people with cognitive impairment will bring a heavy disease burden, and the social cost is almost the sum of cancer, heart disease and stroke.

AD is an age-related neurodegenerative disorder characterized by a progressive decline in cognitive function and daily living capacity. The amyloid hypothesis of AD suggests that the deposition of A β is an early and inevitable event in AD pathogenesis. This hypothesis suggests that therapies that slow the deposition of A β plaques in the brain or increase the clearance of A β may slow the progression of the AD clinical syndrome. Most of the disease course of patients with cognitive impairment is more than 10 years long. How to diagnose and treat them in the early stage has become a key link to delay the progression of the disease and reduce the burden. The disease progression of AD is divided into three major stages: preclinical AD (Preclinical AD, Pre-AD), AD-derived mild cognitive impairment (Mild cognitive impairment due to AD, MCI-AD) and AD dementia (which can be subdivided into mild, moderate and severe AD). Among them, MCI-AD and mild AD are collectively known as early AD, which are the earliest clinical symptoms and the best window for identification and intervention. Studies show that about 43.4% of patients with MCI-AD will progress to AD dementia within 4 years, and 80% will progress within 6 years. If the disease advances to moderate or severe AD, patients will develop severe cognitive, functional impairment and behavioral symptoms, which interfere with social function and need help from daily living activities; severe or even complete loss of independence, requiring round-the-clock care. If early diagnosis and effective interventions in the early stages of the disease, it will help delay the disease into the moderate and severe stages, prolong the quality of life of patients, and greatly reduce the social burden of care and treatment.

At present, the treatment of AD is mainly symptomatic treatment, mainly including cholinesterase inhibitors and NMDA receptor antagonists. Phase-phase clinical trials show that luncinelizumab has a positive impact on cognitive function and pathological indicators in patients with early AD, delaying the early AD disease process by up to 27% relative to placebo treatment. Lencanizumab, a disease-modifying therapy for early AD, has been approved by FDA and NMPA in China. With the wide clinical application, the clinical efficacy and safety of lencanizumab combined with classical symptomatic therapy have attracted great attention. However, there are still few studies on the clinical characteristics, diagnosis and treatment patterns, efficacy and safety of the combination, and clinical outcomes of patients with early AD in the real world.

Based on this, this study intends to conduct an 18-month multi-center prospective real-world observational cohort study exploring the clinical characteristics, diagnosis and treatment patterns, efficacy and safety of the combination, caregiver and family burden of real-world early AD patients (MCI-AD and mild AD).

DETAILED DESCRIPTION:
This study aims to establish a multicenter prospective real-world observational cohort study covering Northeast China, aiming to explore the clinical efficacy and safety of early AD patients combined with conventional drug therapy (luncainizumab combined with conventional drugs), describe the biomarkers and neuroimaging characteristics of early AD (MCI-AD and mild AD) patients in Northeast China; evaluate the cognitive function, daily living ability and neuropsychiatric symptoms of follow-up early AD patients for 18 months; Vertical investigation of family economic burden, caregiver burden, and medical resource utilization in early AD patients in northeast China. It further describes the clinical characteristics, diagnosis and treatment patterns, and the changes of related health outcomes in northeast China in the real world clinical diagnosis and treatment environment.

This study is an 18-month multicenter real-world observational cohort study of 120 early AD patients (MCI-AD and mild AD) attending at 6 centers from January to June 2025, completed the first annual visit from July to December 2025, the second annual visit from January to June 2026, and the third annual visit from July to December 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 50 and 85 years old, male or female;
2. The subjects had primary school education (education) or above, normal hearing, vision and pronunciation, native tongue is Chinese, and daily language is Mandarin, and were able to complete the information collection stipulated in the program.
3. The AD diagnosis met the diagnostic criteria for dementia described in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-R), using the 2011 NIA-AA AD diagnostic criteria. The MCI diagnosis met the MCI diagnostic criteria of Peterson in 2004;
4. The presence of amyloid deposits was confirmed by biomarkers: imaging or cerebrospinal fluid biomarkers.
5. Having cognitive decline, having one of the following conditions: (a) MMSE score of 20 or above; (b) CDR-GS score of 0.5 or 1;
6. The combination group met the criteria for cainumab (according to cainumab instructions);
7. Willing and able to complete all the requirements of the study (including MRI, neuropsychological assessment, clinical genotyping, etc.);
8. Established caregivers or family members can objectively conduct CDR, quality of life scale, daily life performance scale and other clinical assessments;
9. The patient and their family members were informed and signed the informed consent form.

Exclusion Criteria:

1. There are other neurological diseases that can cause brain dysfunction (such as depression, brain tumors, Parkinson's disease, metabolic encephalopathy, encephalitis, multiple sclerosis, epilepsy, brain trauma, normal skull pressure hydrocephalus, etc.);
2. There are other systemic diseases that can cause cognitive impairment (such as liver insufficiency, renal insufficiency, thyroid dysfunction, severe anemia, folic acid or vitamin B12 deficiency, syphilis, HIV infection, alcohol and drug abuse, etc.);
3. Presence of serious or unstable diseases, including cardiovascular, hepatic, renal, gastrointestinal, respiratory, endocrine, neurological (except AD), psychiatric, immune, or hematological diseases and other diseases that the investigator believes may affect the results of the study analysis, or a life expectancy of <24 months;
4. History of schizophrenia, schiztive disorder, major depression or bipolar disorder, and history of major depression may be enrolled in the study if no episodes occurred or mitigated or controlled in the past year; risk of suicide; a history of alcoholism and / or substance abuse or dependence in the past 2 years (according to the Diagnostic and Statistical Manual of Mental Disorders, Version 5th standard)
5. Severe stroke sequelae (mRS> 3 or previous stroke history);
6. Clinically significant systemic immune participants due to the sustained effects of immunosuppressive drugs;
7. Failure to tolerate MRI tests or with MRI contraindications, including but not limited to: a pacemaker incompatible with MRI, eye, skin, MRI clips, artificial heart valve, ear implant, or external metal implant, or other clinical history or findings of which MRI may cause potential harm;
8. Subjects with a history of allergy to any treatment component such as cincainizumab;
9. Refusal to sign the informed consent form.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2025 to June 2025, 120 patients with early AD (MCI-AD and mild AD) who met the inclusion and exclusion criteria and were confirmed to have amyloid protein deposition by biomarkers were selected from 10 centers. Among them, 60 patients were treated with lecanemab combined with symptomatic medication, and the other 60 patients were treated with conventional symptomatic medication.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy and safety of conventional symptomatic drugs combined with lencanizumab in the treatment of early Alzheimer's disease | After collecting the medical information of each follow-up period, the measurement and analysis results will be measured and analyzed.
  Statistical difference in CDR and CDR-SB scores from baseline at 6,12 and 18 months, and in the incidence of adverse reaction events between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Huayan Liu, Study Chair — the first affiliated hospital of China medical university, neurology department

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make IPD and related data dictionaries available.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: starting 12 months after publication
Access Criteria: the IPD and any additional supporting information will be shared with the researchers who follow our idea and theory, and concern on the Efficacy and safety of conventional symptomatic drugs combined with lencanizumab in the treatment of early Alzheimer's disease:. Huayan Liu will review the requests.

REFERENCES:
- [Background] van Dyck CH, Swanson CJ, Aisen P, Bateman RJ, Chen C, Gee M, Kanekiyo M, Li D, Reyderman L, Cohen S, Froelich L, Katayama S, Sabbagh M, Vellas B, Watson D, Dhadda S, Irizarry M, Kramer LD, Iwatsubo T. Lecanemab in Early Alzheimer's Disease. N Engl J Med. 2023 Jan 5;388(1):9-21. doi: 10.1056/NEJMoa2212948. Epub 2022 Nov 29. PMID 36449413
- [Background] Porsteinsson AP, Isaacson RS, Knox S, Sabbagh MN, Rubino I. Diagnosis of Early Alzheimer's Disease: Clinical Practice in 2021. J Prev Alzheimers Dis. 2021;8(3):371-386. doi: 10.14283/jpad.2021.23. PMID 34101796
- [Background] Davis M, O Connell T, Johnson S, Cline S, Merikle E, Martenyi F, Simpson K. Estimating Alzheimer's Disease Progression Rates from Normal Cognition Through Mild Cognitive Impairment and Stages of Dementia. Curr Alzheimer Res. 2018;15(8):777-788. doi: 10.2174/1567205015666180119092427. PMID 29357799
- [Background] Cho SH, Woo S, Kim C, Kim HJ, Jang H, Kim BC, Kim SE, Kim SJ, Kim JP, Jung YH, Lockhart S, Ossenkoppele R, Landau S, Na DL, Weiner M, Kim S, Seo SW. Disease progression modelling from preclinical Alzheimer's disease (AD) to AD dementia. Sci Rep. 2021 Feb 18;11(1):4168. doi: 10.1038/s41598-021-83585-3. PMID 33603015
- [Background] Cohen S, Cummings J, Knox S, Potashman M, Harrison J. Clinical Trial Endpoints and Their Clinical Meaningfulness in Early Stages of Alzheimer's Disease. J Prev Alzheimers Dis. 2022;9(3):507-522. doi: 10.14283/jpad.2022.41. PMID 35841252
- [Background] 王雪莹，李明，卢志明. 阿尔茨海默病生物标志物应用指南及研究进展. 中华预防医学杂志,2022,56(3):262-269.
- [Background] Jia L, Du Y, Chu L, Zhang Z, Li F, Lyu D, Li Y, Li Y, Zhu M, Jiao H, Song Y, Shi Y, Zhang H, Gong M, Wei C, Tang Y, Fang B, Guo D, Wang F, Zhou A, Chu C, Zuo X, Yu Y, Yuan Q, Wang W, Li F, Shi S, Yang H, Zhou C, Liao Z, Lv Y, Li Y, Kan M, Zhao H, Wang S, Yang S, Li H, Liu Z, Wang Q, Qin W, Jia J; COAST Group. Prevalence, risk factors, and management of dementia and mild cognitive impairment in adults aged 60 years or older in China: a cross-sectional study. Lancet Public Health. 2020 Dec;5(12):e661-e671. doi: 10.1016/S2468-2667(20)30185-7. PMID 33271079